CLINICAL TRIAL: NCT02830477
Title: A Multinational Phase IV Study Evaluating "Real World" Treatment Pattern in Previously Treated Hemophilia A Patients Receiving KOVALTRY (Octocog Alfa) for Routine Prophylaxis
Brief Title: Study Evaluating "Real World" Treatment Pattern in Previously Treated Hemophilia A Patients Receiving KOVALTRY (Octocog Alfa) for Routine Prophylaxis
Acronym: TAURUS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18559; KV1601 (Other: Company Internal)
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hemophilia A, Congenital
Keywords: Previously treated patients
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAY81-8973: Previously treated patients receiving IV infusion of KOVALTRY for routine prophylaxis
  Interventions: Biological: Kovaltry (Antihemophilic Factor [Recombinant], BAY81-8973

INTERVENTIONS:
Biological: Kovaltry (Antihemophilic Factor [Recombinant], BAY81-8973 — unmodified, full length recombinant FVIII

SUMMARY:
The primary objective of this study is to investigate weekly prophylaxis dosing regimens used in standard clinical practice.

In addition the study will capture reported bleed rate, pattern of change in KOVALTRY prophylaxis dose & dosing frequency, reason for choice of treatment regimen, FVIII product switch pattern, patient treatment satisfaction and adherence, KOVALTRY pharmacokinetic data (if performed), KOVALTRY consumption, as well as safety data.

DETAILED DESCRIPTION:
Open label, prospective, non-interventional, single arm study in patients receiving KOVALTRY as prophylaxis therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients diagnosed with moderate to severe hemophilia A (≤ 5% FVIII:C (Factor VIII Coagulant activity))
* Any age
* ≥ 50 exposure days (EDs) to any FVIII product
* Patients with or without history of inhibitors

  * Patient with previous history of inhibitors, with at least 2 consecutive negative inhibitor tests and on standard prophylaxis therapy for at least 1 year prior to study entry
  * No current evidence of FVIII inhibitor or clinical suspicion of FVIII inhibitor

    * Evidence of FVIII inhibitor as measured by the Nijmegen-modified Bethesda assay [<0.6 Bethesda units (BU/mL)] or Bethesda assay [< 1.0 BU/mL] in 2 on consecutives samples
    * Documented or clinical suspicion of shortened FVIII half-life (< 6 hrs)
* Currently on or plan to start prophylaxis therapy with KOVALTRY
* Written informed consent

Exclusion Criteria:

* Patients participating in an investigational program with interventions outside of routine clinical practice
* Patients with an additional diagnosis of any bleeding/coagulation disorder other than hemophilia A
* Patients on Immune Tolerance Induction (ITI) treatment at the time of enrollment

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously treated male patients with moderate to severe (≤ 5% FVIII:C) hemophilia A, with ≥ 50 exposure days (EDs) to any FVIII product and with or without history of inhibitors who have been prescribed KOVALTRY for a medically appropriate use will be eligible to be included into this study.
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on 2x and 3x weekly prophylaxis at end of observation period | Up to 2 years

SECONDARY OUTCOMES:
Annualized composite number of reported bleeds (total, spontaneous, joint and trauma) | Up to 2 years
Proportion of patients in predefined prophylaxis regimen per age group and per country | At the end of observational period, up to 2 years
  Age group: 0 to <6, ≥6 to <12, ≥12 to <18, 18 and above
  Weekly prophylaxis dosing regimens:
  * 2 injections a week
  * 3 injections a week
  * Injected on every other day
Physician decision determinants of prophylaxis regimen | At baseline
  Age i.v. access Current treatment regimen Bleeding history with current treatment regimen Prior history of life threatening bleed Number of target joints Pharmacokinetic data Adherence/Compliance history Activity level Patient/caregiver preference Caregiver support Insurance coverage (US) Institution guidelines Country guidelines Other
Change from baseline to one year and two years in treatment satisfaction (Hemo-SAT) | At baseline, 1 year and end of observational period, up to 2 years
  Hemo-SAT - Hemophilia treatment satisfaction questionnaire
Change from baseline to six months, one year and two years in Validated Hemophilia Regimen Treatment Adherence Scale-Prophylaxis (VERITAS-PRO) | At baseline, 6 months and end of observational period, up to 2 years
  VERITAS - Validated Hemophilia Regimen Treatment Adherence Scale-Prophylaxis
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 2 years
Type of data relating to KOVALTRY PK | At routine visits, up to 2 years
  Pharmacokinectic (PK) parameters
  * Area under the curve (AUC)
  * Clearance (Cl)
  * Half-life
  * FVIII trough
  * FVIII peak levels
  * In-vivo recovery
The total annualized factor consumption (injections) | Up to 2 years
Change in prophylaxis dosing frequency (study start to end of observation period) | At baseline and end of observation period, up to 2 years
Reasons for selection of initial dose / dosing frequency of Kovaltry (study start to end of observation period) | At baseline and end of observation period, up to 2 years
Number of KOVALTRY PK assessments performed | At routine visits, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- United States (13):
  - Children's Rehabilitation Services/ University of South Alabama, Mobile, Alabama
  - University of Colorado Hemophilia and Thrombosis Center, Aurora, Colorado
  - University of Florida Health Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic - Division of Pediatric Hematology/Oncology - Jacksonsville, Jacksonville, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Henry Ford Hospital Adult Hemophilia and Thrombosis Treatment Center, Detroit, Michigan
  - Washington University Center for Bleeding and Blood Clotting Disorders, St Louis, Missouri
  - Hemophilia Center of Western New York, Buffalo, New York
  - East Carolina University - Brody School of Medicine, Greenville, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Children's Hospital at OU Medical Center, Oklahoma City, Oklahoma
  - Intermountain Hemophilia & Thrombosis Center, Salt Lake City, Utah
  - Comprehensive Center for Bleeding Disorders / Blood Center of Wisconsin, Milwaukee, Wisconsin
- Multiple Locations, Belgium
- Multiple Locations, Canada
- Multiple Locations, Colombia
- Multiple Locations, France
- Multiple Locations, Germany
- Multiple Locations, Greece
- Multiple Locations, Italy
- Multiple Locations, Luxembourg
- Multiple Locations, Netherlands
- Multiple Locations, Slovenia
- Multiple Locations, Spain
- Multiple Locations, Taiwan

REFERENCES:
- [Result] Santoro C, Fuh B, Le PQ, Maes P, Berrueco R, Mingot-Castellano EM, von Mackensen S, Tueckmantel C, Cabre-Marquez JF, Wang M. Efficacy and safety in patients with haemophilia A switching to octocog alfa (BAY 81-8973): Final results of the global real-world study, TAURUS. Eur J Haematol. 2023 Jan;110(1):77-87. doi: 10.1111/ejh.13876. Epub 2022 Oct 17. PMID 36192847